CLINICAL TRIAL: NCT00364819
Title: Effects of Rituximab (Rituxan) on B Cell and AMA Response in Patients With Primary Biliary Cirrhosis
Brief Title: Initial Study of Rituximab to Treat Primary Biliary Cirrhosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Merrill Eric Gershwin, MD, Principal Investigator, University of California, Davis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200614025
Record Dates: First submitted 2006-08-15; First posted 2006-08-16 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Primary Biliary Cirrhosis
Keywords: Primary Biliary Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): rituximab 1000 mg IV on days 1 and 15, given over 5 - 6 hours
  Interventions: Drug: rituximab

INTERVENTIONS:
Drug: rituximab — rituximab 1000 mg IV day 1 and 15, given over 5 - 6 hours
  Other Names: Rituxan (R)

SUMMARY:
The purpose of this study is to determine the safety of the anti-CD20 antibody rituximab in treating patients with Primary Biliary Cirrhosis (PBC). Rituximab is a laboratory-made antibody currently used to treat some kinds of lymphoma. Rituximab may also help people with PBC, a disease of the immune system. However, the safety of rituximab in PBC patients must first be established.

DETAILED DESCRIPTION:
This is a pilot, open-label, study on 10 female patients with AMA-positive PBC to determine the effects of two infusions of rituximab on response of memory B cells to bacterial motifs, on biochemical function, and histological features. We will enroll 10 consecutive AMA-positive patients with the diagnosis of PBC based on internationally accepted criteria and histological staging determined at liver biopsy and being currently treated with UDCA. Importantly, patients with advanced histological stages, decompensated liver disease, or waiting for OLT will not be included in the study (see exclusion criteria).

Patients eligible and willing to enter the study will be evaluated at baseline by isolation and study of frequency and absolute numbers of B cells and their function, biochemical and AMA tests. Histology and quality of life will be also evaluated in all patients. The methodology to be used for B cell study is already well-established in our laboratory as can be seen in the attached paper (Kikuchi et al. 2005b). Patients will be administered 1,000 mg rituximab intravenously by slow infusion on Day 1 and Day 15 (+/- 1 day). Rituximab's pharmacokinetics indicate that complete B cell depletion is obtained 2-3 days after administration and that such effect may be lost after 9 months (Vieira et al. 2004). In addition to our B cell work, serum samples will undergo AMA testing, including titers, using recombinant mitochondrial antigens (Miyakawa et al. 2001). Patients will also undergo serum chemistry panel, which includes liver function tests. Patients will continue on a steady dose of UDCA therapy throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Liver biopsy showing histological PBC stages I, II, or III
* Presence of all criteria for the diagnosis of PBC
* serum AMA at titer >1:40
* alkaline phosphatase >2X normal value for >6 months
* compatible liver histology
* Incomplete response to UDCA after 6 months of treatment.
* Negative pregnancy test (female patients in fertile age)
* Adequate renal function (serum creatinine < 1.2)

Exclusion Criteria:

* End-stage/decompensated liver disease
* ascites
* jaundice with serum bilirubin > 2mg/dl
* history of digestive bleeding secondary to portal hypertension or endoscopic evidence of varices at stage F2
* history of hepatic encephalopathy
* INR>1.2
* Other coexisting causes of liver disease
* Use of other immunosuppressive medications 4 weeks prior to enrollment
* Diuretics use

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-01; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Eric Gershwin, MD, Principal Investigator — University of California, Davis; Christopher L Bowlus, MD, Study Director — University of California, Davis
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD may be shared upon request and appropriate approval from Institutional Review Boards and material transfer agreements. No patient identifiers will be shared. Requests for IPD may be made to the Principle Investigator.

REFERENCES:
- See also: American Liver Foundation — http://www.liverfoundation.org
- See also: Primary Biliary Cirrhosis Organization — http://www.pbcers.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label Study Arm: Primary Biliary Cirrhosis
  rituximab: rituximab 1000 mg IV day 1 and 15, given over 5 - 6 hours
Period: Overall Study
Arm/Group | Open Label Study Arm
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Open Label Study Arm
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Anti-mitochondrial Antibody [Count of Participants; unit: Participants] — Serum anti-mitochondrial antibodies (AMA) are present in 90% of cases of PBC.
  Participants
    Anti-mitochondrial Antibody Positive | 6
    Anti-mitochondrial Antibody Negative | 0
Liver Biopsy Stage [Count of Participants; unit: Participants] — Staging of liver histology by Ludwig from earliest stage (I) to latest stage (IV). Stage I: Portal inflammation, bile duct abnormalities, or both are present; Stage II: Periportal fibrosis is present, with or without periportal inflammation or prominent enlargement of the portal tracts with seemingly intact, newly formed limiting plates; Stage III: Septal fibrosis with active inflammatory, passive paucicellular septa, or both are present; Stage IV: Nodules with various degrees of inflammation are present
  Participants
    Ludwig Stage I | 1
    Ludwig Stage II | 4
    Ludwig Stage III | 1
    Ludwig Stage IV | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Study Arm
Number analyzed (Participants) | 6
Participants
  Serious Adverse Events | 1
  Non-Serious Adverse Events | 3
  No Events | 2

2. Secondary Outcome: Change in Serum Immunoglobulin G
Description: The difference in serum immunoglobulin G from Baseline to Week 52
Time Frame: 52 Weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Open Label Study Arm
Number analyzed (Participants) | 6
mg/dL | 167 (450)

3. Secondary Outcome: Change in Serum Immunoglobulin A
Description: The difference in serum immunoglobulin A from Baseline to Week 52
Time Frame: 52 Weeks
Population: 1 subject with missing data.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Open Label Study Arm
Number analyzed (Participants) | 5
mg/dL | 36.8 (89.7)

4. Secondary Outcome: Change in Serum Immunoglobulin M
Description: The difference in serum immunoglobulin M from Baseline to Week 52
Time Frame: 52 Weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Open Label Study Arm
Number analyzed (Participants) | 6
mg/dL | 121 (74.5)

5. Secondary Outcome: Change in Serum Alkaline Phosphatase
Description: The difference in serum alkaline phosphatase from Baseline to Week 52
Time Frame: 52 Weeks
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Open Label Study Arm
Number analyzed (Participants) | 6
U/L | 55.8 (151.5)

ADVERSE EVENTS:
Time Frame: 52 weeks after initial infusion of rituximab
Arm/Group | Open Label Study Arm
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Study Arm (N=6)
Shingles (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Study Arm (N=6)
Lymphopenia (Immune system disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No